CLINICAL TRIAL: NCT01972334
Title: A Randomized, Placebo-controlled Pilot Trial to Administer Fecal Microbial Therapy (Stool Transplant) or Placebo in Children Ages 8 to 18 With Recurrent C. Difficile Infection
Brief Title: Stool Transplant in Pediatric Patients With Recurring C. Difficile Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MemorialCare Health System (Other)
Collaborators: Memorial Medical Center Foundation (Other)
Responsible Party: Principal Investigator, Sonia Michail, MD, MD, MemorialCare Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 093-12
Record Dates: First submitted 2013-10-18; First posted 2013-10-30 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Clostridium Difficile Colitis
Keywords: clostridium difficile; children; fecal transplant
MeSH Terms: conditions — Enterocolitis, Pseudomembranous | interventions — Fecal Microbiota Transplantation; Sodium Chloride; Fluoridation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FMT or fecal microbial transplant (Experimental): intervention is fecal microbial transplant done through endoscopy, subjects will be randomized 1:1 to receive either FMT or placebo
  Interventions: Biological: FMT
- placebo (Placebo Comparator): 1:1 randomization to FMT versus placebo (which is saline or salt water)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: FMT — as explained in study arm
  Other Names: fecal microbial transplant; stool transplant
  Arms: FMT or fecal microbial transplant
Biological: placebo — salt water or saline will be given as placebo
  Other Names: saline; salt water
  Arms: placebo

SUMMARY:
The incidence of C. difficile infection (CDI) has alarmingly increased over the past several years and the affected population has expanded to include those previously at low risk, such as children. The annual US financial burden associated with this infection is great and estimated to exceed $1.8 billion. C. difficile infection arises when the gut microbial ecology is disrupted during interventions notorious for perturbing the delicate microbial balance. A well known and common example is the use of antibiotics. Fecal microbiota transplant (FMT) has been introduced several decades ago in an attempt to restore the gut microbial balance. To this date there have been a great number of reports of success in eliminating recurrent C. difficile infections and restoring the gut microbial profile to resemble that of the healthy donor. While over 300 cases have been described in the literature, there has been no pediatric controlled studies performed to compare its efficacy to placebo. Therefore, there is a strong need to determine their safety and efficacy in pediatric randomized controlled studies. The investigators hypothesize that children with recurrent C. difficile infection will respond to fecal transplant therapy which will modify their gut microbial profile. The investigators propose a randomized, placebo controlled, pilot study of fecal microbial transplant in children with recurrent C. difficile infection to evaluate the safety and efficacy of fecal microbial transplant in children in preventing recurrent C. difficile infection. The investigators anticipate that fecal microbial transplant in children with recurrent C. difficile infection will be safe and efficacious and will provide these children with a great alternative to a disease that is difficult to treat. Results of this study will establish the major role of the gut microbiome in this disease and demonstrate the viability of gut microbial transplant in recipients.

DETAILED DESCRIPTION:
Forty six children with recurrent C. difficle infection will be randomized 1:1 to receive either fecal microbial transplant or placebo. The safety and efficacy of this intervention will be monitored for one year.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 1-21.
2. Recurrent C. difficile infection defined as the occurrence of more than two infections

Exclusion Criteria:

1. Inflammatory bowel disease
2. Immune-deficiency.
3. Allergy to oral vancomycin.
4. Children colonized with Clostridium difficile without evidence of symptoms to suggest colitis such as diarrhea and/or rectal bleeding.
5. Concurrent infections that require anti-microbial therapy.
6. Unable to give informed consent/assent.
7. Pregnancy.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome of this randomized, controlled, double-blinded study is the time of recurrence of an infection | 12 months
  secondary outcome measures are focused on the safety of Fecal microbial transplant in this population and all subjects will be closely monitored for developing adverse events for 12 months

SECONDARY OUTCOMES:
safety of fecal microbial transplant in children with recurrent clostridium difficile | 12 months
  All subjects will be closely monitored for adverse events for 12 months after fecal transplant. Subjects will be asked to report any adverse events as they occur and will also be monitored during each visits especially fever, bloating, abdominal pain, vomiting, diarrhea, and rectal bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Michail, MD, Principal Investigator — MemorialCare Health Servies
Locations (1):
- Miller Children's Hospital, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided